CLINICAL TRIAL: NCT02399384
Title: Myocardial Adipose Inflammation and Pericardial Adipose Volume as Markers for Coronary Artery Disease In HIV Positive Patients
Brief Title: Pericardial Fat and Inflammation in HIV Patients and Controls
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, David Harris, Cardiac Imaging Director, University of Cincinnati
Other Study IDs: 2014-6352
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease; Human Immunodeficiency Virus (HIV)
Keywords: Cardiac Magnetic Resonance (CMR)
MeSH Terms: conditions — Coronary Artery Disease; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV+/CAD+: HIV+/CAD+
- HIV+/CAD-: HIV+/CAD-
- HIV-/CAD+: HIV-/CAD+

SUMMARY:
The investigators propose to correlate 1) cardiac MRI pericardial adipose volume, 2) the presence of pericardial monocytes and 3) circulating immune biomarkers in persons with and without CHD and HIV infection compared to seronegative controls with known CHD. The investigators aim to test the hypothesis that higher amounts of pericardial fat deposition and increased presence of monocytes within this adipose tissue are associated with underlying coronary artery disease in persons with HIV infection as measured by cardiac MRI.

DETAILED DESCRIPTION:
Methods and Procedures:

Screening Assessments Patients who potentially meet inclusion criteria will be identified through the Infectious Disease Center and/or the cardiac catheterization laboratory who have had a coronary angiogram or cardiac CT angiogram, with or without evidence of CAD. Their records will be reviewed for inclusion and exclusion criteria and informed consent will be obtained prior to any research related procedures by a member of the research team for this project.

A screening visit will be done to obtain informed consent. BUN and Creatinine will be done at screening to ensure the safety of the MRIprocedure.

In HIV-infected subjects who have not had HIV-1 RNA or CD4+ lymphocyte tests obtained in the last 60 days, these will be done at screening.

Screening visits will last approximately 30-60 minutes.

Entry Visit - MRI The entry visits will occur within 14 days of the screening assessment. All female patients of child bearing potential will have a negative pregnancy test.

If BUN/Creatinine results are greater than 14 days old, they will be repeated STAT prior to beginning MRI procedure.

Whole blood will be drawn for biobanking (PBMCs, Plasma and Serum) as well as fasting lipids will be obtained.

An IV will be started in the MRI laboratory. All participants will undergo an initial cardiac MRI with contrast for the evaluation of cardiac function, chamber size, resting perfusion, pericardial adipose volume/mass, myocardial edema and determination of infarction.

The GE Signa Horizon 1.5T Magnet will be used to obtain all images. Sequences obtained will include Double IR, Triple IR, T2 Stars, SSFP and delayed gadolinium enhancement imaging.

After the initial CMR on day 1, Feraheme 5 mg/kg IV will be administered. Feraheme (30 mg/mL) is available for intravenous injection in single use vials. Each vial contains 510 mg of elemental iron in 17 mL.

Feraheme will be administered as an undiluted intravenous injection delivered at a rate of up to 1 mL/sec (30 mg/sec) through a filtered needle.

Patients will be monitored for 1 hour after administration for signs of allergic reaction.

The total amount of time for the Entry visit will be about 4 hours. Day 2 or 3 - repeat MRI A second, limited cardiac MRI will be obtained 48-72 hours after injection of Feraheme to determine the presence of monocyte/macrophages in adipose tissue.

The GE Signa Horizon 1.5T Magnet will be used to obtain all images. Imaging with T2 Stars and Triple IR sequences.

Data To be Collected:

MRI data to be collected will include:

Left ventricular and right ventricular ejection fractions Left ventricular wall motion Edema Resting myocardial perfusion Pericardial adipose tissue volume T2 star values of pericardial fat pre-Feraheme and post-Feraheme Late gadolinium enhancement (scar assessment and distribution) Valvular assessment Extracardiac assessment - pericardial effusion, pleural effusion, ascites Vital signs (height, weight, blood pressure, heart rate, BSA) Additional Data to be collected if available from the clinical record. Left Heart catheterization Presence or absence of coronary artery disease. The general anatomy, lesion location and severity, presence, location and type of stents, left ventricular end diastolic pressure, systemic blood pressure, aortic valve gradient Echocardiogram Ejection fraction Regional wall motion abnormalities Inducible ischemia if a stress echo was performed Nuclear Stress study Presence or absence of ischemia or infarction Distribution of perfusion abnormalities. Ejection fraction TID (transient ischemic dilatation) End Diastolic Volume End Systolic Volume Medical History (Presence or Absence of ) Sociodemographic information (age, race/ethnicity, etc) HIV related medical information Myocardial Infarction Hypercholesterolemia Hypertension Ventricular Tachycardia Stent Placement Bypass Surgery Diabetes Peripheral Vascular Disease Stroke Smoking (Lifetime Pack-year history and Current status) Family History of Heart Disease Medications Current use in the last 30 days of Anti-hypertensive (Beta Blockers, Calcium Channel Blockers, Ace Inhibitors, Angiotensin Receptor Blockers, Alpha Antagonists) Current use in the last 30 days of Diuretics Lifetime use of Statins Current use in the last 30 days of Insulin or other anti-diabetic medications Lifetime use of Antiretroviral Therapy Laboratory Results HIV-1 Viral Load in the last year Nadir CD4 Count and CD4 count in the last year (include percentages) CD8/CD8 percent in the last year Troponins ( around time of MI if applicable) Most recent Creatinine within 90 days of study entry Most recent BUN within 90 days of study entry If subject has diabetes, hemoglobin A1C or Fructosamine levels in the last year.

Primary endpoints Pericardial adipose tissue volume Change in T2 star value (assessment for iron deposition as a marker for inflammation) Secondary endpoints Correlation of inflammatory biomarkers with Pericardial adipose tissue volume and change in T2 star value Correlation of prior HIV related and Coronary Heart Disease risk factors and events with inflammatory biomarkers, pericardial adipose tissue volume and change in T2 star value.

Data Analysis Data will be stored in a RedCap data base. Statistical analysis will be performed using MedCalc. Continuous variables will be analyzed using analysis of Variance (ANOVA). Non-continuous variables will be analyzed using chi square tests.

Data Monitoring This study will be monitored by a trained coordinator not involved in the research project after enrollment of the first subject, fifth subject and last subject. The monitoring plan will include 100% verification of consent process and inclusion and exclusion criteria. Monitoring for appropriate documentation and collection of study data will be done on the first three subjects and after completion of the last subjects on all study participants. Additional monitoring will be conducted based on risk based assessment of the monitor.

Data Safety Monitoring Board (DSMB) No DSMB will be established for this study. The risks of MRI and phlebotomy are low and there are no test agents being used that are not Food and Drug Administration (FDA) approved. The investigators will monitor closely for adverse events and if an unanticipated number or severity of events occur, the Institutional Review Board (IRB) will be notified and a DSMB will be convened.

Data Storage and Confidentiality:

Participant medical information will be stored electronically in a Redcap database. Each subject will have a unique study ID assigned to their data.

The names and medical record numbers of the research participants will be kept under lock and key and separate from the actual research data in recap. No identifying information will be present in the research database.

Access to participant medical information contained within this research project will be restricted to involved investigators and study personnel.

Password protection of data files will be used. Any paper based data pertaining to individuals will be stored in a locked secure location.

De-identified participant medical record information will be stored for an indefinite period of time per institutional policies at the University of Cincinnati (UC).

Setting: University of Cincinnati Medical Center, and affiliated MRI facilities

Laboratory Methods and Facilities:

Peripheral blood mononuclear cells, plasma and serum will be obtained and stored for subsequent measurement of; hsCRP, IL-6, D-dimer, sCD163, CXCL10, flow cytometry for measures of monocyte activation and additional studies.

DNA will be isolated and may be sent for genetic testing related to inflammation, lipid disorders and atherosclerosis.

Fasting lipids will be obtained on the day of the cardiac MRI CD4 counts and HIV RNA quantitation obtained within 60 days of the cardiac MRI will be recorded.

Estimated Period of Time to Complete the Study: 12 months, ending June 30, 2015.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* History of HIV disease or no history of HIV
* Prior history of left heart catheterization or CTA indicating the presence or absence of CAD.

Exclusion Criteria:

* Unable to have a contrast enhanced cardiac MRI, (i.e. ferromagnetic foreign body, inability to follow verbal instructions, prior history of allergic reactions to gadolinium, history of nephrogenic systemic fibrosis, severe renal dysfunction GFR<30 ml/min/1.73 m2, or severe claustrophobia/anxiety);
* Chronic kidney disease patient undergoing hemodialysis or peritoneal dialysis
* Allergy to Iron Compounds;
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected persons with a history of a positive or negative coronary angiography or cardiac computed tomography angiography (CTA) will be invited to participate in this study from the Infectious Diseases Center practice where there are 1800 persons receiving care. Additionally 4 subjects will be recruited from the cardiology practice at UCMC who have coronary artery disease but do not have HIV.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-01-14 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Pericardial adipose tissue volume | On baseline imaging

SECONDARY OUTCOMES:
Adipose spin spin relaxivity as measured by T2 star time | At baseline and 48-72 hours later

CONTACTS AND LOCATIONS:
Overall Officials: David M Harris, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only researchers approved on the IRB protocol will have access to the data.

REFERENCES:
- [Background] Libby P, Ridker PM, Hansson GK; Leducq Transatlantic Network on Atherothrombosis. Inflammation in atherosclerosis: from pathophysiology to practice. J Am Coll Cardiol. 2009 Dec 1;54(23):2129-38. doi: 10.1016/j.jacc.2009.09.009. PMID 19942084
- [Background] Martinez E, Tuset M, Milinkovic A, Miro JM, Gatell JM. Management of dyslipidaemia in HIV-infected patients receiving antiretroviral therapy. Antivir Ther. 2004 Oct;9(5):649-63. PMID 15535403
- [Background] Paton P, Tabib A, Loire R, Tete R. Coronary artery lesions and human immunodeficiency virus infection. Res Virol. 1993 May-Jun;144(3):225-31. doi: 10.1016/s0923-2516(06)80033-6. PMID 8356344
- [Background] Tabib A, Greenland T, Mercier I, Loire R, Mornex JF. Coronary lesions in young HIV-positive subjects at necropsy. Lancet. 1992 Sep 19;340(8821):730. doi: 10.1016/0140-6736(92)92270-p. No abstract available. PMID 1355828
- [Background] Triant VA, Lee H, Hadigan C, Grinspoon SK. Increased acute myocardial infarction rates and cardiovascular risk factors among patients with human immunodeficiency virus disease. J Clin Endocrinol Metab. 2007 Jul;92(7):2506-12. doi: 10.1210/jc.2006-2190. Epub 2007 Apr 24. PMID 17456578
- [Background] Post WS, Budoff M, Kingsley L, Palella FJ Jr, Witt MD, Li X, George RT, Brown TT, Jacobson LP. Associations between HIV infection and subclinical coronary atherosclerosis. Ann Intern Med. 2014 Apr 1;160(7):458-67. doi: 10.7326/M13-1754. PMID 24687069
- [Background] Obel N, Thomsen HF, Kronborg G, Larsen CS, Hildebrandt PR, Sorensen HT, Gerstoft J. Ischemic heart disease in HIV-infected and HIV-uninfected individuals: a population-based cohort study. Clin Infect Dis. 2007 Jun 15;44(12):1625-31. doi: 10.1086/518285. Epub 2007 May 10. PMID 17516408
- [Background] Triant VA, Meigs JB, Grinspoon SK. Association of C-reactive protein and HIV infection with acute myocardial infarction. J Acquir Immune Defic Syndr. 2009 Jul 1;51(3):268-73. doi: 10.1097/QAI.0b013e3181a9992c. PMID 19387353
- [Background] Mangili A, Polak JF, Quach LA, Gerrior J, Wanke CA. Markers of atherosclerosis and inflammation and mortality in patients with HIV infection. Atherosclerosis. 2011 Feb;214(2):468-73. doi: 10.1016/j.atherosclerosis.2010.11.013. Epub 2010 Nov 17. PMID 21130995
- [Background] Coll B, Parra S, Alonso-Villaverde C, Aragones G, Montero M, Camps J, Joven J, Masana L. The role of immunity and inflammation in the progression of atherosclerosis in patients with HIV infection. Stroke. 2007 Sep;38(9):2477-84. doi: 10.1161/STROKEAHA.106.479030. Epub 2007 Aug 2. PMID 17673719
- [Background] Kaplan RC, Kingsley LA, Gange SJ, Benning L, Jacobson LP, Lazar J, Anastos K, Tien PC, Sharrett AR, Hodis HN. Low CD4+ T-cell count as a major atherosclerosis risk factor in HIV-infected women and men. AIDS. 2008 Aug 20;22(13):1615-24. doi: 10.1097/QAD.0b013e328300581d. PMID 18670221
- [Background] Lang S, Mary-Krause M, Simon A, Partisani M, Gilquin J, Cotte L, Boccara F, Costagliola D; French Hospital Database on HIV (FHDH)-ANRS CO4. HIV replication and immune status are independent predictors of the risk of myocardial infarction in HIV-infected individuals. Clin Infect Dis. 2012 Aug;55(4):600-7. doi: 10.1093/cid/cis489. Epub 2012 May 18. PMID 22610928
- [Background] Choi AI, Li Y, Deeks SG, Grunfeld C, Volberding PA, Shlipak MG. Association between kidney function and albuminuria with cardiovascular events in HIV-infected persons. Circulation. 2010 Feb 9;121(5):651-8. doi: 10.1161/CIRCULATIONAHA.109.898585. Epub 2010 Jan 25. PMID 20100969
- [Background] Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Mateu S, Law M, El-Sadr W, De Wit S, Sabin CA, Phillips AN, Lundgren JD; DAD study group. Cardiovascular disease risk factors in HIV patients--association with antiretroviral therapy. Results from the DAD study. AIDS. 2003 May 23;17(8):1179-93. doi: 10.1097/01.aids.0000060358.78202.c1. PMID 12819520
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Lau B, Sharrett AR, Kingsley LA, Post W, Palella FJ, Visscher B, Gange SJ. C-reactive protein is a marker for human immunodeficiency virus disease progression. Arch Intern Med. 2006 Jan 9;166(1):64-70. doi: 10.1001/archinte.166.1.64. PMID 16401812
- [Background] Feldman JG, Goldwasser P, Holman S, DeHovitz J, Minkoff H. C-reactive protein is an independent predictor of mortality in women with HIV-1 infection. J Acquir Immune Defic Syndr. 2003 Feb 1;32(2):210-4. doi: 10.1097/00126334-200302010-00014. PMID 12571532
- [Background] Ridker PM, Morrow DA, Rose LM, Rifai N, Cannon CP, Braunwald E. Relative efficacy of atorvastatin 80 mg and pravastatin 40 mg in achieving the dual goals of low-density lipoprotein cholesterol <70 mg/dl and C-reactive protein <2 mg/l: an analysis of the PROVE-IT TIMI-22 trial. J Am Coll Cardiol. 2005 May 17;45(10):1644-8. doi: 10.1016/j.jacc.2005.02.080. Epub 2005 Apr 25. PMID 15893181
- [Background] Lowe GD, Rumley A, McMahon AD, Ford I, O'Reilly DS, Packard CJ; West of Scotland Coronary Prevention Study Group. Interleukin-6, fibrin D-dimer, and coagulation factors VII and XIIa in prediction of coronary heart disease. Arterioscler Thromb Vasc Biol. 2004 Aug;24(8):1529-34. doi: 10.1161/01.ATV.0000135995.39488.6c. Epub 2004 Jun 17. PMID 15205218
- [Background] Lowe GD, Sweetnam PM, Yarnell JW, Rumley A, Rumley C, Bainton D, Ben-Shlomo Y. C-reactive protein, fibrin D-dimer, and risk of ischemic heart disease: the Caerphilly and Speedwell studies. Arterioscler Thromb Vasc Biol. 2004 Oct;24(10):1957-62. doi: 10.1161/01.ATV.0000141842.27810.a9. Epub 2004 Aug 12. PMID 15308549
- [Background] Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Neuhaus J, Nixon D, Paton NI, Neaton JD; INSIGHT SMART Study Group. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med. 2008 Oct 21;5(10):e203. doi: 10.1371/journal.pmed.0050203. PMID 18942885
- [Background] Park IW, Wang JF, Groopman JE. HIV-1 Tat promotes monocyte chemoattractant protein-1 secretion followed by transmigration of monocytes. Blood. 2001 Jan 15;97(2):352-8. doi: 10.1182/blood.v97.2.352. PMID 11154208
- [Background] Fisher SD, Miller TL, Lipshultz SE. Impact of HIV and highly active antiretroviral therapy on leukocyte adhesion molecules, arterial inflammation, dyslipidemia, and atherosclerosis. Atherosclerosis. 2006 Mar;185(1):1-11. doi: 10.1016/j.atherosclerosis.2005.09.025. Epub 2005 Nov 16. PMID 16297390
- [Background] Burdo TH, Lo J, Abbara S, Wei J, DeLelys ME, Preffer F, Rosenberg ES, Williams KC, Grinspoon S. Soluble CD163, a novel marker of activated macrophages, is elevated and associated with noncalcified coronary plaque in HIV-infected patients. J Infect Dis. 2011 Oct 15;204(8):1227-36. doi: 10.1093/infdis/jir520. PMID 21917896
- [Background] Sani MU. Myocardial disease in human immunodeficiency virus (HIV) infection: a review. Wien Klin Wochenschr. 2008;120(3-4):77-87. doi: 10.1007/s00508-008-0935-3. PMID 18322768
- [Background] Raj V, Joshi S, Pennell DJ. Images in Cardiovascular Medicine. Cardiac magnetic resonance of acute myocarditis in an human immunodeficiency virus patient presenting with acute chest pain syndrome. Circulation. 2010 Jun 29;121(25):2777-9. doi: 10.1161/CIRCULATIONAHA.109.888099. No abstract available. PMID 20585023
- [Background] Restrepo CS, Diethelm L, Lemos JA, Velasquez E, Ovella TA, Martinez S, Carrillo J, Lemos DF. Cardiovascular complications of human immunodeficiency virus infection. Radiographics. 2006 Jan-Feb;26(1):213-31. doi: 10.1148/rg.261055058. PMID 16418253
- [Background] Konishi M, Sugiyama S, Sugamura K, Nozaki T, Ohba K, Matsubara J, Matsuzawa Y, Sumida H, Nagayoshi Y, Nakaura T, Awai K, Yamashita Y, Jinnouchi H, Matsui K, Kimura K, Umemura S, Ogawa H. Association of pericardial fat accumulation rather than abdominal obesity with coronary atherosclerotic plaque formation in patients with suspected coronary artery disease. Atherosclerosis. 2010 Apr;209(2):573-8. doi: 10.1016/j.atherosclerosis.2009.10.008. Epub 2009 Oct 12. PMID 19892354
- [Background] de Vos AM, Prokop M, Roos CJ, Meijs MF, van der Schouw YT, Rutten A, Gorter PM, Cramer MJ, Doevendans PA, Rensing BJ, Bartelink ML, Velthuis BK, Mosterd A, Bots ML. Peri-coronary epicardial adipose tissue is related to cardiovascular risk factors and coronary artery calcification in post-menopausal women. Eur Heart J. 2008 Mar;29(6):777-83. doi: 10.1093/eurheartj/ehm564. Epub 2007 Dec 20. PMID 18156138
- [Background] Katsiki N, Mikhailidis DP, Wierzbicki AS. Epicardial fat and vascular risk: a narrative review. Curr Opin Cardiol. 2013 Jul;28(4):458-63. doi: 10.1097/HCO.0b013e3283605fba. PMID 23591557
- [Background] Gronemeyer SA, Steen RG, Kauffman WM, Reddick WE, Glass JO. Fast adipose tissue (FAT) assessment by MRI. Magn Reson Imaging. 2000 Sep;18(7):815-8. doi: 10.1016/s0730-725x(00)00168-5. PMID 11027874
- [Background] Machann J, Thamer C, Schnoedt B, Haap M, Haring HU, Claussen CD, Stumvoll M, Fritsche A, Schick F. Standardized assessment of whole body adipose tissue topography by MRI. J Magn Reson Imaging. 2005 Apr;21(4):455-62. doi: 10.1002/jmri.20292. PMID 15778954
- [Background] Nelson AJ, Worthley MI, Psaltis PJ, Carbone A, Dundon BK, Duncan RF, Piantadosi C, Lau DH, Sanders P, Wittert GA, Worthley SG. Validation of cardiovascular magnetic resonance assessment of pericardial adipose tissue volume. J Cardiovasc Magn Reson. 2009 May 5;11(1):15. doi: 10.1186/1532-429X-11-15. PMID 19416534
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Rajiah P. Cardiac MRI: Part 2, pericardial diseases. AJR Am J Roentgenol. 2011 Oct;197(4):W621-34. doi: 10.2214/AJR.10.7265. PMID 21940533
- [Background] Weinsaft JW, Kim HW, Shah DJ, Klem I, Crowley AL, Brosnan R, James OG, Patel MR, Heitner J, Parker M, Velazquez EJ, Steenbergen C, Judd RM, Kim RJ. Detection of left ventricular thrombus by delayed-enhancement cardiovascular magnetic resonance prevalence and markers in patients with systolic dysfunction. J Am Coll Cardiol. 2008 Jul 8;52(2):148-57. doi: 10.1016/j.jacc.2008.03.041. PMID 18598895
- [Background] Schelbert EB, Cao JJ, Sigurdsson S, Aspelund T, Kellman P, Aletras AH, Dyke CK, Thorgeirsson G, Eiriksdottir G, Launer LJ, Gudnason V, Harris TB, Arai AE. Prevalence and prognosis of unrecognized myocardial infarction determined by cardiac magnetic resonance in older adults. JAMA. 2012 Sep 5;308(9):890-6. doi: 10.1001/2012.jama.11089. PMID 22948699
- [Background] Greenwood JP, Maredia N, Younger JF, Brown JM, Nixon J, Everett CC, Bijsterveld P, Ridgway JP, Radjenovic A, Dickinson CJ, Ball SG, Plein S. Cardiovascular magnetic resonance and single-photon emission computed tomography for diagnosis of coronary heart disease (CE-MARC): a prospective trial. Lancet. 2012 Feb 4;379(9814):453-60. doi: 10.1016/S0140-6736(11)61335-4. Epub 2011 Dec 22. PMID 22196944
- [Background] Kellman P, Aletras AH, Mancini C, McVeigh ER, Arai AE. T2-prepared SSFP improves diagnostic confidence in edema imaging in acute myocardial infarction compared to turbo spin echo. Magn Reson Med. 2007 May;57(5):891-7. doi: 10.1002/mrm.21215. PMID 17457880
- [Background] Kellman P, Arai AE. Imaging sequences for first pass perfusion --a review. J Cardiovasc Magn Reson. 2007;9(3):525-37. doi: 10.1080/10976640601187604. PMID 17365232
- [Background] Schelbert EB, Hsu LY, Anderson SA, Mohanty BD, Karim SM, Kellman P, Aletras AH, Arai AE. Late gadolinium-enhancement cardiac magnetic resonance identifies postinfarction myocardial fibrosis and the border zone at the near cellular level in ex vivo rat heart. Circ Cardiovasc Imaging. 2010 Nov;3(6):743-52. doi: 10.1161/CIRCIMAGING.108.835793. Epub 2010 Sep 16. PMID 20847191
- [Background] Iles L, Pfluger H, Phrommintikul A, Cherayath J, Aksit P, Gupta SN, Kaye DM, Taylor AJ. Evaluation of diffuse myocardial fibrosis in heart failure with cardiac magnetic resonance contrast-enhanced T1 mapping. J Am Coll Cardiol. 2008 Nov 4;52(19):1574-80. doi: 10.1016/j.jacc.2008.06.049. PMID 19007595
- [Background] Arai AE. The cardiac magnetic resonance (CMR) approach to assessing myocardial viability. J Nucl Cardiol. 2011 Dec;18(6):1095-102. doi: 10.1007/s12350-011-9441-5. PMID 21882082
- [Background] Sandstede J, Lipke C, Beer M, Hofmann S, Pabst T, Kenn W, Neubauer S, Hahn D. Age- and gender-specific differences in left and right ventricular cardiac function and mass determined by cine magnetic resonance imaging. Eur Radiol. 2000;10(3):438-42. doi: 10.1007/s003300050072. PMID 10756992
- [Background] Haddad F, Hunt SA, Rosenthal DN, Murphy DJ. Right ventricular function in cardiovascular disease, part I: Anatomy, physiology, aging, and functional assessment of the right ventricle. Circulation. 2008 Mar 18;117(11):1436-48. doi: 10.1161/CIRCULATIONAHA.107.653576. No abstract available. PMID 18347220
- [Background] Grothues F, Moon JC, Bellenger NG, Smith GS, Klein HU, Pennell DJ. Interstudy reproducibility of right ventricular volumes, function, and mass with cardiovascular magnetic resonance. Am Heart J. 2004 Feb;147(2):218-23. doi: 10.1016/j.ahj.2003.10.005. PMID 14760316
- [Background] Weissleder R, Stark DD, Engelstad BL, Bacon BR, Compton CC, White DL, Jacobs P, Lewis J. Superparamagnetic iron oxide: pharmacokinetics and toxicity. AJR Am J Roentgenol. 1989 Jan;152(1):167-73. doi: 10.2214/ajr.152.1.167. PMID 2783272
- [Background] Wang YX, Hussain SM, Krestin GP. Superparamagnetic iron oxide contrast agents: physicochemical characteristics and applications in MR imaging. Eur Radiol. 2001;11(11):2319-31. doi: 10.1007/s003300100908. PMID 11702180
- [Background] Chapon C, Franconi F, Lemaire L, Marescaux L, Legras P, Saint-Andre JP, Denizot B, Le Jeune JJ. High field magnetic resonance imaging evaluation of superparamagnetic iron oxide nanoparticles in a permanent rat myocardial infarction. Invest Radiol. 2003 Mar;38(3):141-6. doi: 10.1097/01.RLI.0000052979.96332.90. PMID 12595793
- [Background] Sosnovik DE, Nahrendorf M, Deliolanis N, Novikov M, Aikawa E, Josephson L, Rosenzweig A, Weissleder R, Ntziachristos V. Fluorescence tomography and magnetic resonance imaging of myocardial macrophage infiltration in infarcted myocardium in vivo. Circulation. 2007 Mar 20;115(11):1384-91. doi: 10.1161/CIRCULATIONAHA.106.663351. Epub 2007 Mar 5. PMID 17339546
- [Background] Ho C, Hitchens TK. A non-invasive approach to detecting organ rejection by MRI: monitoring the accumulation of immune cells at the transplanted organ. Curr Pharm Biotechnol. 2004 Dec;5(6):551-66. doi: 10.2174/1389201043376535. PMID 15579044
- [Background] Oweida AJ, Dunn EA, Foster PJ. Cellular imaging at 1.5 T: detecting cells in neuroinflammation using active labeling with superparamagnetic iron oxide. Mol Imaging. 2004 Apr;3(2):85-95. doi: 10.1162/15353500200404106. PMID 15296673
- [Background] Rausch M, Hiestand P, Baumann D, Cannet C, Rudin M. MRI-based monitoring of inflammation and tissue damage in acute and chronic relapsing EAE. Magn Reson Med. 2003 Aug;50(2):309-14. doi: 10.1002/mrm.10541. PMID 12876707
- [Background] Pennell DJ, Sechtem UP, Higgins CB, Manning WJ, Pohost GM, Rademakers FE, van Rossum AC, Shaw LJ, Yucel EK; European Society of cardiology; Soceity for Cardiovascular Magnetic Resonance. Clinical indications for cardiovascular magnetic resonance (CMR): Consensus Panel report. J Cardiovasc Magn Reson. 2004;6(4):727-65. doi: 10.1081/jcmr-200038581. No abstract available. PMID 15646878